CLINICAL TRIAL: NCT01263080
Title: Multicentre Randomised Double-blind, Placebo-controlled 2x2 Factorial Trial Investigating the Effects of Adding Mirtazapine and Folic Acid to Existing Therapy for Patients With Schizophrenia
Brief Title: Evaluation of Mirtazapine and Folic Acid for Schizophrenia:
Acronym: RECOVERY2
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Capital Medical University (Other)
Responsible Party: Principal Investigator, Gang Wang, vice-director of Affective Disorder Center, Beijing Anding Hospital, Capital Medical University
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: RECOVERY2
Record Dates: First submitted 2010-12-17; First posted 2010-12-20 (Estimated); Last update posted 2016-08-02 (Estimated); Status verified 2016-08

CONDITIONS: Schizophrenia
Keywords: mirtazapine; folic acid; schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — Mirtazapine; Folic Acid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- mirtazapine+folic acid (Active Comparator): mirtazapine 30mg QD, folic acid 0.4mg QD
  Interventions: Drug: mirtazapine; Drug: folic acid
- mirtazapine+folic acid placebo (Active Comparator): mirtazapine 30mg QD, folic acid placebo 1 tablet QD
  Interventions: Drug: mirtazapine; Drug: folic acid placebo
- mirtazapine placebo+folic acid (Active Comparator): mirtazapine placebo 1 tablet QD, folic acid 0.4mg QD
  Interventions: Drug: mirtazapine placebo; Drug: folic acid
- mirtazapine placebo+folic acid placebo (Placebo Comparator): mirtazapine placebo 1 tablet QD, folic acid placebo 1 tablet QD
  Interventions: Drug: folic acid placebo; Drug: mirtazapine placebo

INTERVENTIONS:
Drug: mirtazapine — mirtazapine 30mg QD
  Other Names: Remeron
  Arms: mirtazapine+folic acid; mirtazapine+folic acid placebo
Drug: folic acid placebo — folic acid placebo 1 tablet QD
  Other Names: Folic placebo
  Arms: mirtazapine placebo+folic acid placebo; mirtazapine+folic acid placebo
Drug: mirtazapine placebo — mirtazapine placebo 1 tablet QD
  Other Names: Remeron placebo
  Arms: mirtazapine placebo+folic acid; mirtazapine placebo+folic acid placebo
Drug: folic acid — folic acid 0.4mg QD
  Other Names: vitamin B 9
  Arms: mirtazapine placebo+folic acid; mirtazapine+folic acid

SUMMARY:
Multicentre randomised double-blind, placebo-controlled 2x2 factorial trial investigating the effects of adding mirtazapine and folic acid to existing therapy for patients with schizophrenia

DETAILED DESCRIPTION:
The combination of mirtazapine plus antipsychotic potentially offers considerable benefit for patients with schizophrenia. Folic acid is a promising adjunctive therapy for schizophrenia that may also provide benefits for patients with other mental disorders. Furthermore the effects of folic acid may be affected by genotype.

The trial will investigate the effects of adding mirtazapine and the effects of adding folic acid to treatments for schizophrenia. At randomisation, patients will be separately randomised to mirtazapine or placebo and to folic acid or placebo.

Randomised, double-blind, placebo-controlled 2x2 factorial trial with 12-week follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Inpatients or outpatients age 18 to 70 years;
2. Meet DSM-IV criteria for schizophrenia;
3. Signed an informed consent form by patients or their legally acceptable representatives;
4. PANSS total score >=60 and at least one item of P1, P2, P3, P5 or P6 >=4 to ensure subject has current active psychotic symptoms - i.e. hallucinations, delusions, thought disorder;
5. Subjects who are currently taking effective dose of antipsychotic;
6. Women must agree to practice an effective method of birth control if they are sexually active before entry and throughout the study.

Exclusion Criteria:

1. Meet any other DSM-IV Axis I disorders;
2. Meet DSM-IV criteria for substance abuse or dependence;
3. Have been treatment-resistant to 2 or more kinds of antipsychotics with sufficient dosage for at least 4 weeks, or require clozapine treatment, or have received clozapine treatment within 1 month prior to randomization;
4. Subjects are actively suicidal or judged clinically to be at risk of serious suicidal or violent behavior in the opinion of the investigator;
5. Have serious or unstable medical illness (e.g., cardiovascular disease, neurologic, hematologic, renal, hepatic, immunologic, endocrine, or other systemic illness), or have any clinically significant abnormality on laboratory test or ECG which indicate severe medical conditions;
6. Have received electroconvulsive therapy within 28 days before randomization;
7. Have received long acting antipsychotic within 1 treatment cycle before randomization;
8. Have received antidepressant within 14 days, or have received MAOIs within 4 weeks before randomization or require antidepressive treatment;
9. History of prostatic hypertrophy or dysuria;
10. History of narrow-angle glaucoma or elevation of intraocular pressure;
11. Known or suspected history of allergy or have contradiction to mirtazapine or folic acid;
12. Known have currently requirement of taking mirtazapine or folic acid;
13. Women who are pregnant or nursing;
14. Have previously completed or withdrawn from this study, or participated in a clinical trial of another drug within 30 days.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 333 (Actual)
Dates: Start 2010-11; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
To compare the efficacy of mirtazapine and placebo for treatment of symptoms associated with schizophrenia | baseline, week4, week8, week12

SECONDARY OUTCOMES:
To compare the efficacy of folic acid and placebo for treatment of symptoms of schizophrenia | baseline, week4, week8, week12
To compare the efficacy of mirtazapine and placebo for treatment of negative symptoms of schizophrenia | baseline, week4, week8, week12
To compare the efficacy of folic acid and placebo for treatment of negative symptoms of schizophrenia | baseline, week4, week8, week12
To compare the safety and tolerability of mirtazapine and placebo in patients with schizophrenia | baseline, week4, week8, week12
To compare the safety and tolerability of folic acid and placebo in patients with schizophrenia | baseline, week4, week8, week12

CONTACTS AND LOCATIONS:
Overall Officials: Gang Wang, M.D., Principal Investigator — Beijing Anding Hospital, Capital Medical University
Locations (1):
- Beijing Anding Hospital, Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided